CLINICAL TRIAL: NCT04793425
Title: The Impact of Mobile Application and a Digital Support System on the Prevention of Cardiovascular Events in Patients After a Myocardial Infarction.
Brief Title: Mobile App and Digital System for Patients After Myocardial Infarction
Acronym: afterAMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WarsawMU1
Record Dates: First submitted 2021-02-04; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2020-12

CONDITIONS: mHealth; Telemedicine
Keywords: Myocardial infarction; Telemedicine; Mobile health
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Patients randomized to standard care arm will take part in the rehabilitation program according to regular schedule. Additionally every patient will have 2 cardiological visits: 1 and 6 months after the hospitalization due to MI.
- Mobile app care (Experimental): Patients randomized to standard care arm will take part in the rehabilitation program according to regular schedule. Additionally every patient will have 2 cardiological visits: 1 and 6 months after the hospitalization due to MI. On top of that every patient will be given an access to mobile application, which will support rehab process. The application stands as a educational and coordination tool.
  Interventions: Behavioral: Mobile application (afterAMI)

INTERVENTIONS:
Behavioral: Mobile application (afterAMI) — The rehabilitation process of the patients in the intervention group will be supported by the mobile application (afterAMI) with synchronized, dedicated web page.
  Patients in the intervention group will be given an access to educational data regarding their individualized diseases. Additionally every patient will receive regularly messages with notifications regarding lifestyle and adherence to the therapy. All reported vital signs (blood pressure, heart rate, weight and many more) will be analyzed every day and in case of need a short message will be sent to the patient with indication to go to the primary healthcare clinic/hospital.
  Additionally, application will send notifications with reminders to take drugs.
  Arms: Mobile app care

SUMMARY:
The treatment of acute myocardial infarction (MI) in Poland is at the level of standardized European care. However, the first months after MI are crucial from the perspective of patient's prognosis. It is extremely important to take care of all cardiovascular risk factors.

Mobile application (afterAMI) supported by web system is a novel telemedical tool created to support patient and physician during the process of cardiac rehabilitation. The application has educational model with focus on cardiovascular risk factors and lifestyle after MI. Moreover, there is a module to control vital signs like blood pressure, heart rate, weight and many others. Additionally, application will send reminders for better drug adherence.

100 patients will be recruited to take part in the study. All of which will be hospitalized at the 1st Department and Clinic of Cardiology because of the MI. The aim of the project is to study the impact of application-supported model of care with comparison to standard care. At the end of the study cardiovascular risk factors control will be analysed, as well as rehospitalizations, patient's knowledge regarding risk factors, return to work and quality of life.

This will be a prospective, open-label, randomized, single-centre study. All 100 patients will be observed 6 months after discharge from the hospital. End points will be assessed during control visit 1- and 6-months after inclusion into the study.

This project is an example of a telemedicine solution application into everyday practice, which is consistent with multiple international cardiac societies.

ELIGIBILITY:
Inclusion Criteria:

* signing the informed consent to participate in the study
* hospitalization due to myocardial infarction
* a mobile device with Internet access and the Android/iOS operating system
* age >17 years old
* positive results of the test verifying the basic skills of using mobile applications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Rehospitalization or urgent outpatient visit | This outcome will be assessed 1 month after discharge from the hospital.
  The number and reasons of rehospitalizations and urgent outpatient visits.
Rehospitalization or urgent outpatient visit | This outcome will be assessed 6 months after discharge from the hospital.
  The number and reasons of rehospitalizations and urgent outpatient visits.
Cardiovascular risk factors control - hypertension | This outcome will be assessed 1 month after discharge from the hospital.
  Systolic and diastolic blood pressure values will be analyzed with special focus on meeting the values recommended by European Society of Cardiology guidelines.
Cardiovascular risk factors control - hypertension | This outcome will be assessed 6 months after discharge from the hospital.
  Systolic and diastolic blood pressure values will be analyzed with special focus on meeting the values recommended by European Society of Cardiology guidelines.
Cardiovascular risk factors control - body mass | This outcome will be assessed 1 month after discharge from the hospital.
  Body mass will be measured. Change [kg] from baseline body mass will be analyzed.
Cardiovascular risk factors control - body mass | This outcome will be assessed 6 months after discharge from the hospital.
  Body mass will be measured. Change [kg] from baseline body mass will be analyzed.
Cardiovascular risk factors control - nicotinism | This outcome will be assessed 1 month after discharge from the hospital.
  The number of patients who are active smokers will be assessed. The change from baseline will be analyzed.
Cardiovascular risk factors control - nicotinism | This outcome will be assessed 6 months after discharge from the hospital.
  The number of patients who are active smokers will be assessed. The change from baseline will be analyzed.
Cardiovascular risk factors control - dyslipidemia | This outcome will be assessed 1 month after discharge from the hospital.
  LDL cholesterol level will be measured and the change from baseline will be analyzed.
Cardiovascular risk factors control - dyslipidemia | This outcome will be assessed 6 months after discharge from the hospital.
  LDL cholesterol level will be measured and the change from baseline will be analyzed.

SECONDARY OUTCOMES:
Quality of life - MacNew | This outcome will be assessed 1 month after discharge from the hospital.
  Quality of life will be assessed with MacNew questionnaire.Scoring of the MacNew is straight-forward. The maximum possible score in any domain is 7 [high quality] and the minimum is 1 [poor quality]. The quality of life is assessed with regard to physical, emotional and social aspect, as well as general quality of life. There are 27 questions in total.
Quality of life - MacNew | This outcome will be assessed 6 months after discharge from the hospital.
  Quality of life will be assessed with MacNew questionnaire.Scoring of the MacNew is straight-forward. The maximum possible score in any domain is 7 [high quality] and the minimum is 1 [poor quality]. The quality of life is assessed with regard to physical, emotional and social aspect, as well as general quality of life. There are 27 questions in total.
Quality of life - descriptive profile of a respondent's health state | This outcome will be assessed 1 month after discharge from the hospital.
  Quality of life will be assessed with EQ-5D-5L questionnaire. The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group.
  There are 5 aspects examined: mobility, self-care, usual activity, pain/discomfort, anxiety/depression. Every part is assessed based on 5 level scale:
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems
Quality of life - descriptive profile of a respondent's health state | This outcome will be assessed 6 months after discharge from the hospital.
  Quality of life will be assessed with EQ-5D-5L questionnaire. The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group.
  There are 5 aspects examined: mobility, self-care, usual activity, pain/discomfort, anxiety/depression. Every part is assessed based on 5 level scale:
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems
DASS 21 - Depression, anxiety and stress assessment | This outcome will be assessed 1 month after discharge from the hospital.
  Depression, anxiety and stress assessment will be assessed with DASS 21 (Depression Anxiety Stress Scales) scale The DASS is a quantitative measure of distress along the 3 axes of depression, anxiety and stress.
  There are 21 questions, each has 4 possible answers:
  0 Did not apply to me at all - NEVER
  1. Applied to me to some degree, or some of the time - SOMETIMES
  2. Applied to me to a considerable degree, or a good part of time - OFTEN
  3. Applied to me very much, or most of the time - ALMOST ALWAYS There are 7 questions assigned to every aspect: depression, anxiety and stress respectively.
  Higher result in every section contributes to higher severity in depression, anxiety and stress.
DASS 21 - Depression, anxiety and stress assessment | This outcome will be assessed 6 months after discharge from the hospital.
  Depression, anxiety and stress assessment will be assessed with DASS 21 (Depression Anxiety Stress Scales) scale The DASS is a quantitative measure of distress along the 3 axes of depression, anxiety and stress.
  There are 21 questions, each has 4 possible answers:
  0 Did not apply to me at all - NEVER
  1. Applied to me to some degree, or some of the time - SOMETIMES
  2. Applied to me to a considerable degree, or a good part of time - OFTEN
  3. Applied to me very much, or most of the time - ALMOST ALWAYS There are 7 questions assigned to every aspect: depression, anxiety and stress respectively.
  Higher result in every section contributes to higher severity in depression, anxiety and stress.
  Higher result in every section contributes to higher severity in depression, anxiety and stress.
Cardiovascular risk factor knowledge | This outcome will be assessed 1 month after discharge from the hospital.
  Cardiovascular risk factor knowledge will be assessed with previously prepared questionnaire (10 questions).
  There are 9 single choice questions. Every correct answer is rewarded with a point. There is 1 open question, where the patient is asked to list known cardiovascular risk factors. Patient gets 1 point fo 1-2 CV risk factors, 2 points for 3-4 CV risk factors, 3 points for 5-6 CV risk factors and 4 points for >6 named CV risk factors.
  The maximum score is 13 points , which indicates good cardiovascular risk factors knowledge. The minimum score is 0 points, which indicates poor cardiovascular risk factors knowledge.
Cardiovascular risk factor knowledge | This outcome will be assessed 6 months after discharge from the hospital.
  Cardiovascular risk factor knowledge will be assessed with previously prepared questionnaire (10 questions).
  There are 9 single choice questions. Every correct answer is rewarded with a point. There is 1 open question, where the patient is asked to list known cardiovascular risk factors. Patient gets 1 point fo 1-2 CV risk factors, 2 points for 3-4 CV risk factors, 3 points for 5-6 CV risk factors and 4 points for >6 named CV risk factors.
  The maximum score is 13 points , which indicates good cardiovascular risk factors knowledge. The minimum score is 0 points, which indicates poor cardiovascular risk factors knowledge.
Return to work | This outcome will be assessed 1 month after discharge from the hospital.
  In case of patients who were previously working the amount of patients who came back to work will be assessed.
Return to work | This outcome will be assessed 6 months after discharge from the hospital.
  In case of patients who were previously working the amount of patients who came back to work will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Department of Cariology of Medcial University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krzowski B, Peller M, Boszko M, Hoffman P, Zurawska N, Jaruga K, Skoczylas K, Osak G, Koltowski L, Grabowski M, Opolski G, Balsam P. Mobile app and digital system for patients after myocardial infarction (afterAMI): study protocol for a randomized controlled trial. Trials. 2022 Jun 21;23(1):522. doi: 10.1186/s13063-022-06463-x. PMID 35729626